CLINICAL TRIAL: NCT02834611
Title: Phase I Study of C6 Ceramide NanoLiposome in Patients With Advanced Solid Tumors
Brief Title: Ceramide NanoLiposome in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Keystone Nano, Inc (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KNAN1001; R44CA195793 (NIH)
Record Dates: First submitted 2016-07-11; First posted 2016-07-15 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Cancer; Carcinoma; Solid Tumors; Tumor
MeSH Terms: conditions — Neoplasms; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ceramide NanoLiposome (Experimental): Dose escalation of Ceramide NanoLiposome
  Interventions: Drug: Ceramide NanoLiposome

INTERVENTIONS:
Drug: Ceramide NanoLiposome — Intravenous administration of Ceramide NanoLiposome

SUMMARY:
This study is a dose escalation study of Ceramide NanoLiposome in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent/authorization is obtained prior to conducting any study-specific screening procedures.
* 18 years of age or order
* Histologic or cytologic diagnosis of cancer
* Patients without a curative therapy or whose tumor does not have standard chemotherapy
* At least 4 weeks after the last dose of chemotherapy or radiation therapy; 6 weeks for mitoxantrone or mitomycin therapy
* Eastern Cooperative Oncology Group (ECOG) performance status must be ≤2 (Appendix A).
* Adequate hepatic, renal, and bone marrow function:

  * Absolute neutrophil count ≥ 1,000/microliter (uL)
  * Platelets ≥ 100,000/uL
  * Total bilirubin ≤2.0
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional ULN
  * Creatinine ≤1.2 mg/dL or clearance ≥50ml/min (Cockcroft-Gault)
* All participants (male and female) with reproductive potential must practice an effective method of contraception while on this study in order to minimize risks to fetuses.
* Radiographic evidence of measurable disease tumor lesion (≥ 1cm in greatest dimension) or nodal disease (>1.5cm in greatest dimension)
* Men and women of all ethnic groups are eligible for this trial.
* Females at reproductive age must have a negative urine pregnancy test prior to entry to this study
* Life expectancy is greater than 12 weeks.
* Patients with controlled CNS disease and off steroids are eligible.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmias not well controlled with medication, myocardial infarction within the previous 6 months, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients may not be receiving any other concurrent investigational agents, or have received any investigational agent within four weeks of commencing this protocol.
* Since the teratogenic potential of this combination is currently unknown, females who are pregnant or lactating are excluded. Males and females should perform abstinence or use barrier to prevent pregnancy.
* History of any other malignancies in the last 2 years except in-situ cancer, non-muscle invasive bladder cancer, basal or squamous cell skin cancer are eligible
* Patients known to be HIV(+), Hep BsAg(+), or Hep C(+) are excluded as the effect of the agent on immune system has not been assessed
* Patients with history of hypersensitivity to liposomal products
* Patients with primary CNS malignancies or leptomeningeal disease are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of Ceramide NanoLiposome in patients with advanced solid tumors. | 24 months

SECONDARY OUTCOMES:
Recommended phase II dose | 24 months
Incidence of treatment-related adverse events as assessed by CTCAE v4.0 | 24 months
Peak plasma concentration (Cmax) | 24 months
Time to maximum plasma concentration (Tmax) | 24 months
Ceramide NanoLiposome half-life (t1/2) | 24 months
Objective response rate per RECIST v1.1 | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward Sausville, MD, PhD, Principal Investigator — University of Maryland Greenebaum Cancer Center
Locations (3):
- United States (3):
  - University of Maryland, Greenebaum Cancer Center, Baltimore, Maryland
  - Medical University of South Carolina, Hollings Cancer Center, Charleston, South Carolina
  - University of Virginia Cancer Center, Charlottesville, Virginia

REFERENCES:
- [Derived] Ciner A, Gourdin T, Davidson J, Parette M, Walker SJ, Fox TE, Jiang Y. A phase I study of the ceramide nanoliposome in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2024 Jan;93(1):23-29. doi: 10.1007/s00280-023-04588-7. Epub 2023 Sep 22. PMID 37736793